CLINICAL TRIAL: NCT04293991
Title: High Flow Nasal Cannula Versus Non Invasive Ventilation in Prevention of Intubbation in Immunocompromised Patient With Acute Hypoxxemic Respiratory Failure
Brief Title: High Flow Nasal Cannula in Immunocompromised Patient With Acute Respiratory Failure
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Ain Shams University (Other)
Responsible Party: Principal Investigator, Ashraf Elsayed Elagamy, Assisstant professor Anesthesia,Intensive care and pain management, Ain Shams University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: FMASU R 9 / 2020
Record Dates: First submitted 2020-02-22; First posted 2020-03-03 (Actual); Last update posted 2020-03-03 (Actual); Status verified 2020-02

CONDITIONS: High Flow Nasal Cannula; Non Invasive Ventilation; Acute Respiratory Failure
Keywords: High flow nasal cannula, .; Non invasive ventilation
MeSH Terms: interventions — Noninvasive Ventilation

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- High flow nasal cannula (HFNC) group (Active Comparator): HFNC group will receive immediate connection to HFNC with a flow of 60L/min, and FIO2 adjusted to have SpO2 of 92% or more, through a heated humidifier and a oxygen blender of the same machine. In case of patient intolerance to high flow, flow will be diminished to the highest tolerated by the patient. Patients will be encouraged to have their mouth closed during HFNC to augment positive end expiratory pressure (PEEP) created by high flow.
  Interventions: Device: High Flow Nasal Cannula
- Non invasive ventilation (NIV) group (Active Comparator): NIV group, patients will be connected to ICU ventilatoron NIV mode for at least 4 hours, through a NIV continuous positive airway pressure (CPAP)mask with ventilator settings; pressure support (PS) level of 8 cmH2O and PEEP level of 5 cmH2O,which can be increased to 10 cmH2O to maintain tidal volume between 6-8 ml/Kg and FiO2 adjusted to keep SpO2 equal or more than 92%.At least patient will be on NIV for 12 hours during the day, alternating with Venturi mask 10-15 L/min to keep FiO2 equal or more than 92%.
  Interventions: Device: Non Invasive Ventilation

INTERVENTIONS:
Device: High Flow Nasal Cannula — Evaluate the use of HFNC in prevention of intubation in immunocompromised patients adimitted to icu.
  Arms: High flow nasal cannula (HFNC) group
Device: Non Invasive Ventilation — Evaluate the use of HFNC in prevention of intubation in immunocompromised patient admitted to icu.
  Arms: Non invasive ventilation (NIV) group

SUMMARY:
This study will be conducted in Ain Shams University Hospital in the general intensive care unit after ethical committee approval number (FMASU R 9/2020) .It is a prospective randomized controlled study. Eligible patients will be randomized by computer system to one of two groups either High Flow Nasal Oxygen (HFNO) group or Non Invasive Ventilation (NIV) group. Inclusion criteria includes admitted immunocompromised patients to our general 34 beds ICU with acute hypoxemic respiratory failure (ARF).

DETAILED DESCRIPTION:
ARF is characterized by respiratory rate more than 25/min, PaO2/FiO2 less than 300 under standard O2 10 L/min, or findings of persistent pulmonary infiltrates in radiographs.

Immunocompromised patients have one or more of the following criteria hematological malignancy (either active or remitting in the last 5 years), bone marrow transplantation (in the last 5 years), severe leucopenia less than 1000 white blood cells in cubic millimeter, solid organ transplantation, steroid therapy more than 0.5 mg/kg/day for at least 3 weeks, or cytotoxic therapy for non malignant disease.

Patients included in the study will be randomized after admission to ICU to one of two groups, HFNC group or NIV group. Patients enrolled in HFNC group will receive immediate connection to HFNC with a flow of 60L/min, and FIO2 adjusted to have SpO2 of 92% or more, through a heated humidifier and a oxygen blender of the same machine. In case of patient intolerance to high flow, flow will be diminished to the highest tolerated by the patient. Patients will be encouraged to have their mouth closed during HFNC to augment positive end expiratory pressure (PEEP) created by high flow.NIV group, patients will be connected to ICU ventilator on NIV mode for at least 4 hours, through a NIV continuous positive airway pressure (CPAP)mask with ventilator settings; pressure support (PS) level of 8 cmH2O and PEEP level of 5 cmH2O,which can be increased to 10 cmH2O

ELIGIBILITY:
Inclusion Criteria:

* . Inclusion criteria includes admitted immunocompromised patient to ICU with acute hypoxemic respiratory failure (ARF).
* Hematological malignancies.
* Post bone marrow transplantation

Exclusion Criteria:

* Need of emergency intubation.
* patient with deterioration of conscious level with hypoxemia with FiO2 less than 90% in spite of maximum O2 support.

  * hemodynamic instability with need of vasoconstrictor support.

Ages: 18 Years to 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 76 (Estimated)
Dates: Start 2020-03 (Estimated); Primary Completion 2020-07 (Estimated); Study Completion 2020-08 (Estimated)

PRIMARY OUTCOMES:
primary outcome will be need for endotracheal intubation within 48 hours of admission | 48 hours of patient admission to ICU.
  Need for endotracheal intubation within 48 hours of admission to ICU

SECONDARY OUTCOMES:
secondary outcome will be mortality rate after 28 days of admission. | 28 days after patient admission to ICU.
  mortality rate after 28 days after patient admission to ICU.

CONTACTS AND LOCATIONS:
Overall Officials: Sameh Salem, MD, Study Director — Professor Doctor

IPD SHARING:
Plan to Share IPD: No
Not yet decided that patient participating will accept for share their information or no.